CLINICAL TRIAL: NCT02566512
Title: Assessment of Cough Strength in Patients With Tracheostomies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: B2015:068
Record Dates: First submitted 2015-06-23; First posted 2015-10-02 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Mechanical Ventilator Weaning
Keywords: Tracheostomy; weaning; respiratory failure; cough strength
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tracheostomy cuff inflated (Other): The tracheostomy cuff will be inflated.
  Interventions: Other: Tracheostomy cuff inflation.
- Tracheostomy cuff deflated (Other): The tracheostomy cuff will be deflated.
  Interventions: Other: Tracheostomy cuff deflation

INTERVENTIONS:
Other: Tracheostomy cuff inflation. — With the tracheostomy cuff inflated, the peak expiratory flow meter will be attached directly to the tracheostomy tube. The patient will be instructed to take as big a breath as they can and then forcefully cough. This will be repeated four times.
  Arms: Tracheostomy cuff inflated
Other: Tracheostomy cuff deflation — With the tracheostomy cuff deflated, a one-way valve will be attached to the tracheostomy tube. The patient will use a mouthpiece to connect to the peak expiratory flow meter. The patient will be instructed to take as big a breath as they can and then forcefully cough. This will be repeated four times
  Arms: Tracheostomy cuff deflated

SUMMARY:
The investigators propose to assess cough strength in patients undergoing spontaneous breathing trials in the Intermediate Intensive Care Unit (IICU) and compare their cough strength under two conditions,

1. Tracheostomy cuff inflated: cough strength will be measured with the tracheostomy cuff inflated and the patient coughing through the tracheostomy tube.
2. Tracheostomy cuff deflated: cough strength will be measured with the tracheostomy cuff deflated and the patient coughing around the tracheostomy tube, through their mouth..

The investigators hypothesize that patients will have a stronger cough when they can use their vocal cords.

DETAILED DESCRIPTION:
When a patient has recovered from the initial respiratory insult which precipitated respiratory failure, the patient may need a prolonged period of time to wean completely from mechanical ventilation.

One method of weaning from mechanical ventilation involves having the patient breath spontaneously without the assistance of the ventilator. This is referred to as a spontaneous breathing trial. Over time, the duration of spontaneous breathing is gradually increased until the patient is able to breathe entirely on their own. Traditionally, the tracheostomy cuff has been kept inflated until the patient can breathe entirely on their own (2,3).

A recent study has assessed the effect of deflating the tracheostomy tube cuff on weaning from mechanical ventilation (4). Patients, who required prolonged mechanical ventilation and had a tracheostomy, were weaned using a T piece trial. They were randomized to two groups: the control group had the tracheostomy cuff kept inflated; the study group had the tracheostomy cuff deflated. The study group, with the cuff deflated, had a shorter time to weaning from the ventilator, fewer respiratory infections and improved swallowing. This was attributed to an increase in the effective airway diameter, which would decrease the resistive work of breathing. The authors did not comment on the effect cuff deflation may have on coughing and clearance of secretions.

It is postulated that patients can cough more effectively when he/she can use their vocal cords to generate a cough as opposed to coughing through a tracheostomy tube where the vocal cords are bypassed. It has been previously demonstrated that patients have a stronger cough after the tracheostomy tube has been removed as compared to when the tracheostomy tube is in place (5).

Patient population

The study group will include all adult patients in the IICU, on prolonged mechanical ventilation who are having spontaneous breathing trials as part of their weaning protocol.

Patients will be required to give written, informed consent.

Exclusion criteria

Any patient who has a leak around their tracheostomy tube when the tracheostomy cuff is inflated.

Inability to understand English or cognitive impairment which impairs the patient's ability to follow directions.

Protocol

Baseline demographic information will be collected from each patient. This will include age, sex, height, weight, BMI, diagnosis, initial date of intubation and ICU admission, date of tracheostomy, date of admission to IICU, type and size of tracheostomy tube.

Baseline measurements of respiratory strength will be made in all patients. These will include vital capacity (VC), maximal inspiratory pressure (MIP), and maximal expiratory pressure (MEP). These are standard measurements, routinely done in the IICU. All measurements will be done with the patient in a head up or sitting position with the tracheostomy cuff inflated.

Measurement of cough strength will be done using an Air Zone Peak Expiratory Flow meter. This will be done with the patient in a head up or sitting position.

With the tracheostomy cuff inflated, the peak expiratory flow meter will be attached directly to the tracheostomy tube. The patient will be instructed to take as big a breath as they can and then forcefully cough. This will be repeated four times. The first measurement will be discarded (learning curve). The peak expiratory flow will be recorded for the next three measurements. The three measurements should not deviate by more than 10%, and the best result will be recorded.

With the tracheostomy cuff deflated, a one-way valve will be attached to the tracheostomy tube. The patient will use a mouthpiece to connect to the peak expiratory flow meter. The patient will be instructed to take as big a breath as they can and then forcefully cough. This will be repeated four times. The first measurement will be discarded (learning curve). The peak expiratory flow will be recorded for the next three measurements. The three measurements should not deviate by more than 10 %, and the best result will be recorded.

The patients will be randomized to start with either the tracheostomy cuff inflated or deflated.

At the end of the measurements, the patient will be returned to their usual care.

The entire study should take approximately ten minutes.

The investigators propose to study 20 consecutive adult patients in the IICU.

Data analysis

The best expiratory flow measurements will be averaged together with the tracheostomy cuff inflated and with the tracheostomy cuff deflated. The values will be compared using Student's T test. A p value < 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* The study group will include all adult patients in the IICU, on prolonged mechanical ventilation who are having spontaneous breathing trials as part of their weaning protocol.

Exclusion Criteria:

* Any patient who has a leak around their tracheostomy tube when the tracheostomy cuff is inflated.
* Inability to understand English or cognitive impairment which impairs the patient's ability to follow directions.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-09; Primary Completion 2018-09 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Peak expiratory flow rate | Twenty minutes
  peak flow rate during a cough

CONTACTS AND LOCATIONS:
Overall Officials: Eric Jacobsohn, MD, Study Chair — University of Manitoba
Locations (1):
- Health Sciences Centre, Winnipeg, Manitoba, Canada

REFERENCES:
- [Result] Daniel Martin A, Smith BK, Gabrielli A. Mechanical ventilation, diaphragm weakness and weaning: a rehabilitation perspective. Respir Physiol Neurobiol. 2013 Nov 1;189(2):377-83. doi: 10.1016/j.resp.2013.05.012. Epub 2013 May 18. PMID 23692928
- [Result] Frutos-Vivar F, Esteban A. Our paper 20 years later: how has withdrawal from mechanical ventilation changed? Intensive Care Med. 2014 Oct;40(10):1449-59. doi: 10.1007/s00134-014-3362-0. Epub 2014 Jul 23. PMID 25053247
- [Result] Hernandez G, Pedrosa A, Ortiz R, Cruz Accuaroni Mdel M, Cuena R, Vaquero Collado C, Garcia Plaza S, Gonzalez Arenas P, Fernandez R. The effects of increasing effective airway diameter on weaning from mechanical ventilation in tracheostomized patients: a randomized controlled trial. Intensive Care Med. 2013 Jun;39(6):1063-70. doi: 10.1007/s00134-013-2870-7. Epub 2013 Mar 8. PMID 23471512
- [Result] McKim DA, Hendin A, LeBlanc C, King J, Brown CR, Woolnough A. Tracheostomy decannulation and cough peak flows in patients with neuromuscular weakness. Am J Phys Med Rehabil. 2012 Aug;91(8):666-70. doi: 10.1097/PHM.0b013e31825597b8. PMID 22561386
- [Result] Heffner JE, Martin-Harris B. (2006) Care of the Mechanically Ventilated Patient with a Tracheostomy in Tobin MJ (Ed) Principles and Practice of Mechanical Ventilation 2nd edition (pp 847 - 875) McGraw-Hill